CLINICAL TRIAL: NCT00086125
Title: A Phase II Study of AP23573, an mTOR Inhibitor, in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: Study of AP23573 in Patients With Relapsed or Refractory Hematologic Malignancies (8669-024)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-024; AP23573-04-201
Record Dates: First submitted 2004-06-24; First posted 2004-06-28 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Hematologic Malignancies; Leukemia; Myelodysplastic Syndromes; Myeloid Metaplasia; Lymphoma
Keywords: Relapsed or refractory hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma; Recurrence | interventions — ridaforolimus

ARMS (1):
- 1 (Experimental): AP23573 12.5 mg IV as monotherapy once daily for 5 days, every 2 weeks
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — AP23573 12.5 mg IV as monotherapy once daily for 5 days, every 2 weeks
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
The purpose of this phase II study is to assess the efficacy of AP23573 in patients with specified relapsed or refractory hematological malignancies.

DETAILED DESCRIPTION:
The primary objective of the trial is to assess the efficacy of AP23573 in patients with specified relapsed or refractory hematological malignancies by evaluating the response rates as defined for the individual malignancy categories. Secondary objectives include evaluating time to disease progression, progression-free survival and duration of response; evaluating the pharmacokinetic and pharmacodynamic characteristics of AP23573; describing health-related quality of life measurements; and exploring the safety and tolerability of AP23573 at the specified dose level.

Protocol Outline: Open label, non-randomized parallel cohorts of five disease-specific cohorts with a minimum of 21 patients per cohort. Each patient receives a fixed dose of AP23573 administered intravenously (IV) over 30 minutes daily for five days (QDx5) to be repeated every 2 weeks.

ELIGIBILITY:
Inclusion Criteria (Patients must meet each of the following criteria to be eligible for participation in the trial):

* Male or female patients ≥ 18 years of age
* Patients must have histologically-confirmed diagnoses of relapsed or refractory hematologic malignancy as specified in the protocol
* Patients must have an ECOG performance status of 0 to 2
* Patients must have adequate renal and liver function as demonstrated by laboratory values performed within 5 days, inclusive, prior to administration of the first dose of AP23573
* Patients must be able to understand and give written informed consent

Exclusion Criteria (Patients meeting any of the following criteria are ineligible for participation in the study):

* Women who are pregnant or lactating
* Patients may not have had cytotoxic chemotherapy or radiotherapy within 14 days prior to study entry
* Patients may not receive any investigational anti-cancer agent while on this study or within 14 days prior to the first dose of AP23573
* Patients with known or suspected hypersensitivity to drugs formulated with polysorbate 80 (Tween) or any other excipient contained in the study drug formulation
* Patients with known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
* Patients with significant uncontrolled cardiovascular disease
* Patients with known HIV infection
* Patients with any uncontrolled infection
* Patients receiving immunosuppressive agents other than prescribed corticosteroids
* Patients who have had prior therapy with rapamycin, any rapamycin analog or tacrolimus
* Patients with inadequate recovery from any prior surgical procedure or patients having undergone any major surgical procedure within 14 days prior to the first dose of AP23573
* Patients with any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug
* Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies
* Patients with another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinomas in situ)
* Patients with the inability, in the opinion of the Investigator, to comply with the protocol requirements

Drugs and Other Treatments to be Excluded (The following drugs and other treatments are not permitted for patients enrolling in the study, either during or within two weeks prior to the first dose of AP23573, unless otherwise specified):

* Chemotherapeutic agents with the following exception that therapy with nitrosoureas (including generics) cannot be given within six weeks prior to the first dose of AP23573
* Other antineoplastic agents
* Immunotherapy (including vaccines) or biological response modifier therapy
* Systemic hormonal therapy with exceptions as specified in the protocol
* Herbal preparations or related OTC preparations containing herbal ingredients (e.g., St John's Wort)
* Radiotherapy for the primary malignancy
* Any other investigational agent during the course of the trial should be discussed with the Sponsor prior to use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of AP23573 in patients with relapsed or refractory hematologic malignancies. | Duration of study

SECONDARY OUTCOMES:
Evaluating time to progression, progression-free survival, duration of response and safety | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, M.D., Ph.D., Study Director — Ariad Pharmaceuticals
Locations (8):
- United States (8):
  - University of Chicago Hospitals, Section of Hematology/Oncology, Chicago, Illinois
  - Washington University School of Medicine, Siteman Cancer Center, 4921 Parkview Place, St Louis, Missouri
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Presbyterian Hospital, Weill College of Cornell University, New York, New York
  - Morris Cancer Center - Duke University Medical Center, Adult Bone Marrow Transplant Clinic, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Jeane's Hospital of TUHS, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Rizzieri DA, Feldman E, Dipersio JF, Gabrail N, Stock W, Strair R, Rivera VM, Albitar M, Bedrosian CL, Giles FJ. A phase 2 clinical trial of deforolimus (AP23573, MK-8669), a novel mammalian target of rapamycin inhibitor, in patients with relapsed or refractory hematologic malignancies. Clin Cancer Res. 2008 May 1;14(9):2756-62. doi: 10.1158/1078-0432.CCR-07-1372. PMID 18451242